CLINICAL TRIAL: NCT06293521
Title: Clinical and Radiographic Success Rate of Pulpotomy Versus Pulpectomy for Management of Primary Teeth With Deep Caries: A Randomized Clinical Trial
Brief Title: Clinical and Radiographic Success Rate of Pulpotomy Versus Pulpectomy for Management of Primary Teeth With Deep Caries
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nada Mohamed Hassan Mostafa, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06091995
Record Dates: First submitted 2024-02-14; First posted 2024-03-05 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Deep Caries
Keywords: Irreversible pulpits; Pulpotomy; Pulpectomy
MeSH Terms: interventions — Pulpotomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MTA Pulpotomy (Experimental): Intervention group
  Interventions: Procedure: Pulpotomy
- Chlorohexidine Pulpectomy (Active Comparator): Control group
  Interventions: Procedure: Partial Pulpectomy

INTERVENTIONS:
Procedure: Pulpotomy — After the chamber is deroofed and coronal pulp is amputated using a round-end fissure bur in a high-speed handpiece with adequate water spray and light pressure until canal orifices were reached, The access cavity is flushed with sterile normal saline solution. Saline-wetted cotton pellets were placed for about 5 minutes over amputation sites applying moderate pressure to control pulpal hemorrhage. After discarding the pellets, blood oozing was present, MTA+ Cerkamed will be manipulated in the ratio of 3:1 (powder: liquid) to obtain a putty mix. This mix will be placed over the radicular pulp with the help of a suitable sterile amalgam carrier. Gentle condensation of the mix will be done in the pulp chamber with a moistened cotton pellet, followed by application of glass ionomer cement.
  Arms: MTA Pulpotomy
Procedure: Partial Pulpectomy — Pulp tissue extirpation is done. Biomechanical preparation is done using rotary files with frequent irrigation with Chlorhexidine. The canals are dried using sterile absorbent paper points followed by obturation by the paste of Zinc oxide and eugenol.
  The tooth with then be restored with stainless steel crown
  Arms: Chlorohexidine Pulpectomy

SUMMARY:
This trial aims to compare treatment outcomes between Pulpotomy and Pulpectomy in treating vital primary teeth diagnosed with deep caries with symptoms of irreversible pulpits

DETAILED DESCRIPTION:
Background: Pulpectomy is the reference treatment for vital primary molars with irreversible pulpitis.Over the past decades, dental caries has unfailingly been the most common chronic infectious disease of childhood and adults. If remained untreated, it can potentially compromise dental pulp tissue. When the dental pulp of primary teeth is irreversibly inflamed, the first treatment choice is pulpectomy, owing to the well-recognized importance of primary tooth retention for child oral/general health. Although a pulpless tooth can remain functional in the oral cavity, modern pediatric endodontics encourages regenerative approaches in primary teeth.The introduction of calcium silicate-based (CS-B) biomaterials such as mineral trioxide aggregate (MTA), along with further understanding of pulp biology and inflammatory processes, has revolutionized treatment modalities for management of irreversible pulpitis in mature permanent teeth. A growing body of evidence has revealed successful implementation of minimally invasive endodontics, that is, vital pulp therapies (VPTs) for management of permanent teeth with irreversible pulpitis even when associated with apical periodontitis. Due to the traditional notion of poorer healing capacity of primary dental pulp, such a paradigm shift has not been seen in pediatric dentistry.Recent research revealed similar vascular/immune responses of primary and permanent dental pulps to caries; therefore, indicating that their healing potential might be this in mind, a reevaluation of traditional approaches for treatment of inflamed primary pulp seems justified.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 4 to 6 years , in good general health
2. The parents provided written informed consent.
3. Clinical characteristics, defined as spontaneous pain and the presence of a deep carious lesion with pulp exposure and bleeding that did not halt within five minutes following removal of the coronal pulp tissue.
4. Restorable teeth.

Exclusion Criteria:

1. Physical or mental disability.
2. Unable to attend follow-up visits.
3. Previously accessed teeth.
4. Swelling, tenderness to percussion or palpation, or pathological mobility.
5. Pre-operative radiographic pathology such as resorption (internal or external), per-radicular or furcation radiolucency.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic assessment | Month 6 , Month 12
  Absence of periapical radiolucency or absence of internal/ external root resorption

SECONDARY OUTCOMES:
Clinical effectiveness | Month 3,Month 6,Month 9,Month 12
  absence of any complication or complementary treatment: Absence of spontaneous pain & Absence of swelling.
Child cooperation | Day 0
  Modified frankl scale ,Categorical rating (rating 1 is definitly negative
  - Rating 5 is definitely positive )
Time elapsed till final restoration performed | Day 0
  Stopwatch , measured in minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt